CLINICAL TRIAL: NCT05234762
Title: A Phase 2A, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of ES-481 in Adult Patients With Essential Tremors
Brief Title: Efficacy, Safety, and Pharmacokinetics of ES-481 in Adult Patients With Essential Tremors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ES Therapeutics Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ES-481-C203
Record Dates: First submitted 2021-11-27; First posted 2022-02-10 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Tremor, Essential
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES-481 (Experimental): Week 1 - 25 mg qd (2 x 25 mg capsule in the mornings Days 1 to 7 in Treatment Period 1 and Days 44 to 50 in Treatment Period 2) Week 2 - 50 mg bid (2 x 25 mg capsule in the mornings and 2 x 25 mg capsules in the evening on Days 8 to 14 in Treatment Period 1 and Days 51 to 57 in Treatment Period 2) Week 3 - 75 mg bid (2 x 25 mg capsule in the mornings and 2 x 25 mg capsules in the evening on Days 15 to 21 in Treatment Period 1 and Days 58 to 64 in Treatment Period 2) Week 4 - 75 mg bid (2 x 25 mg capsule in the mornings and 2 x 25 mg capsules in the evening on Days 22 to 28 in Treatment Period 1 and Days 65 to 71 in Treatment Period 2)
  Interventions: Drug: ES-481
- Placebo (Placebo Comparator): Placebo will be dosed at the same quantity and frequency as ES-481 just as Placebo HPMC capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ES-481 — Dose escalation during two Treatment Periods
  Arms: ES-481
Other: Placebo — Placebo dosed at same dosing as ES-481
  Arms: Placebo

SUMMARY:
This Pilot Phase 2A study will investigate the safety, tolerability, and pharmacokinetics (PK) of ES-481 in adult patients with essential tremor.

ELIGIBILITY:
Inclusion Criteria:

* Written and Signed Informed Consent
* Age 18 to 75 years old
* The Subject must have Essential Tremor (ET). ET is defined as at least 1 upper extremity with a tremor score ≥ 1.5 in forward posture, wing beating posture, or finger-to-nose movement using the Performance subscale of The Essential Tremor Rating Assessment Scale (as per by the Tremor Investigation Group criteria).
* Subject has a diagnosis of essential tremor, as defined by all the following criteria: (a) isolated tremor syndrome consisting of bilateral upper limb action; (b) at least three years duration; (c) with or without tremor in other location (e.g., head, voice, or lower limb).
* The Subject must be on stable dose of anti-tremor medication in the four (4) weeks prior to screening and must willing to maintain their current dose for the duration of the study.
* The Subject had no prior surgery for tremor.
* The Subject had no botulinum injection for at least six (6) months prior to -screening.
* The Subject does not have a significant imbalance or risk fall.
* The Subject has not previously taken perampanel.

Exclusion Criteria:

Subjects will be excluded from 7-day screening period or study enrollment into the Treatment Period 1, if they meet any of the following criteria:

* Unwilling or inability to follow the procedures specified by the protocol
* Pregnancy or breast feeding
* Women of child-bearing potential and men who are unable or unwilling to take adequate contraceptive precautions, including one of the following:

  * Hormonal contraception (birth control pills, injected hormones, or vaginal ring)
  * Intrauterine device
  * Barrier methods (condom or diaphragm) combined with spermicide
  * Surgical sterilization (hysterectomy, tubal ligation, or vasectomy)
* History (within the last year) of illicit drug use or alcohol dependence or a positive screen for alcohol on the Day 1 visit, or a positive screen for drugs of abuse at Screening or at the Day 1 visit
* Subject is unwilling or unable to refrain from alcohol 24 hours before and during clinical trial visits, or regular use of alcohol that would preclude abstinence from alcohol for time periods around visits.
* Subject has a history of substance use disorder consistent with Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria, in the opinion of the Principal Investigator,
* Concomitant treatment with more than three drugs to treat essential tremors
* Subject has had recent exposure (14 days prior to Day 1) to tremorgenic drugs.
* Subject has had direct or indirect injury or trauma to the nervous system within 3 months before the onset of tremor.
* Subject has a history or clinical evidence of other medical, neurological, or psychiatric conditions that may explain or cause tremors, including but not limited to Parkinson's disease, Huntington's disease, cerebellar disease (including spinocerebellar ataxias, primary dystonia, Fragile X Tremor/Ataxia syndrome or Family history of Fragile X syndrome, traumatic brain injury, psychogenic tremor, alcohol or benzodiazepines abuse or withdrawal, multiple sclerosis, polyneuropathy, and endocrine states such as hyperthyroidism or unstable treatment of hypothyroidism or medication, food, or supplement induced movement disorder (e.g., tremor related to beta agonists or caffeine), or other medical, neurological or psychiatric condition that may explain or cause tremors.
* Subject has had a previous procedure for the treatment of ET, deep brain stimulation, brain lesioning, or magnetic resonance (MR)-guided procedure, e.g., MR-guided focused ultrasound.
* Subject has historical or clinical evidence of tremor with psychogenic origin (including but not limited to eating disorders, major depression, etc.).
* Subject has history of suicidal behavior within 2 years or is currently at risk for suicide in the opinion of the investigator.
* Subject has any neurological abnormality other than ET upon neurological exam, including dystonia, ataxia, or any other neurodegenerative disease, including multiple sclerosis.
* Subject has alkaline phosphatase, aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT) level >3.0 x upper limit of normal (ULN) at Screening and/or at Pre-dose.
* Subject has serum creatinine >120 μmol/L and/or creatinine clearance <60 mL/min (according to Cockcroft-Gault formula) at Screening.
* Subject has a history of Long QT syndrome and/or QTcF (Fridericia's correction) interval >450 msec (males) or >470 msec (females) per 12-lead ECG done at Screening.
* Subject has a diagnosis of epilepsy or any history of seizure as an adult; head trauma, stroke, transient ischemic attack within 1 year prior to Screening; unexplained loss of consciousness within 1 year prior to Screening; or any lifetime history of asymptomatic or symptomatic orthostatic hypotension (e.g., postural syncope)
* Subject has a history of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class 3 or 4), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year prior to screening.
* Subject has any major psychiatric disorder that is uncontrolled (for the past 90 days) that, per the Investigator's judgment, can interfere with any of the study procedures.
* Subject should not have received treatment with another investigational drug within 30 days or 5 half-lives (whichever is longer), prior to the screening visit.
* Subject should not have received a vaccine within 60 days prior to study drug administration, except for vaccines related to Covid-19.
* Subject should not have donated or lost more than 450mL of blood or received a transfusion of any blood or blood products within 90 days prior to screening, or donated plasma within 7 days prior to admission.
* Subject has a known allergy to ES-481 or its excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance Subscale of The Essential Tremor Rating Assessment Scale (TETRAS-P) | Collected during 6 days throughout the study, scores to be combined.
  To evaluate postural and kinetic tremor of body parts affected by ET, with emphasis on upper extremity tremor. Items are scored from 0 to 4, with 4 representing the highest severity.
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Total protein
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Sodium
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Potassium
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Calcium
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Chloride
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Albumin
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Glucose
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Blood urea nitrogen (BUN)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Creatinine
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Carbon dioxide (CO2)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Uric acid
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Total bilirubin
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Alkaline phosphatase (AP)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: AST
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: ALT
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Gamma-glutamyl transpeptidase (GGT)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Lactate dehydrogenase (LDH)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Creatine phosphokinase (CPK)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Hemoglobin
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Hematocrit
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Red blood cell (RBC) count
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: White blood cell (WBC) count with differential
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Mean corpuscular volume (MCV)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Mean corpuscular hemoglobin (MCH)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Mean corpuscular hemoglobin (MCHC)
Number of participants with abnormal laboratory test results | Through study completion, an average of 78 days.
  Collection of: Absolute platelet count
Safety assessments through collection of serious adverse events | Through study completion, an average of 78 days.
  Collection of Serious Adverse Events
Safety assessments through collection of adverse events | Through study completion, an average of 78 days.
  Collection of Adverse Events
Safety assessments through collection of treatment emergent adverse events | Through study completion, an average of 78 days.
  Collection of Treatment Emergent Adverse Events
Plama samples for PK | Will be collected on Days 1, 22, 29, 44, 65, and 72
  Will be collected to assess the plasma concentration of ES-481 during the 28-day treatment periods from both ES-481 and Placebo subjects to estimate the PK of ES-481 After the study blind is broken, only the samples from subjects who took ES-481 will be analyzed.

SECONDARY OUTCOMES:
Activity of Daily Living | Will be completed on Days 1 (baseline and prior to administration of study medication on Day 1 in Treatment Period 1), and Days 22, 29, 44 (baseline and prior to administration of study medication on Day 44 in Treatment Period 2), 65, and 72
  Subjects will complete a 12-item (0-4 ratings) Activity of Daily Living questionnaire.
Subject Global Impression of Change Scale (SGIC) | Will be completed on Days 1 (baseline and prior to administration of study medication on Day 1 in Treatment Period 1), and Days 22, 29, 44 (baseline and prior to administration of study medication on Day 44 in Treatment Period 2), 65, and 72
  Subjects will rate overall change with the Subject Global Impression of Change Scale in which change was rated between minus 3 and plus 3, with 1 connoting mild change, 2 moderate change, and 3 marked changes, with minus indicating improvement and plus worsening

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Neuro-Levis, Lévis, Quebec, Canada